CLINICAL TRIAL: NCT06261489
Title: The Differential Effects of THC vs. CBD on Cognition in Persons With MS
Brief Title: Cannabis (THC vs. CBD) in Multiple Sclerosis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Multiple Sclerosis Society of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB23-1128
Record Dates: First submitted 2024-01-10; First posted 2024-02-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Cannabis; Cognitive Function
MeSH Terms: conditions — Multiple Sclerosis; Marijuana Abuse | interventions — Dronabinol; Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tetrahydrocannabinol (THC) 25 mg (Experimental): THC oil will be administered orally once a day for 15 weeks.
  Interventions: Drug: THC
- Cannabidiol (CBD) 50 mg (Experimental): CBD oil will be administered orally once a day for 15 weeks.
  Interventions: Drug: CBD

INTERVENTIONS:
Drug: THC — Participants will be randomly assigned to the study treatment. THC dose will be gradually increased until 25 mg. Treatment will be taken orally at bedtime for 15 weeks.
  Other Names: Tetrahydrocannabinol
  Arms: Tetrahydrocannabinol (THC) 25 mg
Drug: CBD — Participants will be randomly assigned to the study treatment. CBD dose will be gradually increased until 50 mg. Treatment will be taken orally at bedtime for 15 weeks.
  Other Names: Cannabidiol
  Arms: Cannabidiol (CBD) 50 mg

SUMMARY:
The goal of this clinical trial is to examine the effect of Cannabis components, THC and CBD, on cognition and bladder symptoms in people with Multiple Sclerosis (MS).

Participants will complete questionnaires and cognitive tests. They will be randomly assigned to receive either CBD or THC oil and will take the study drug for 15 weeks.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic autoimmune disease of the central nervous system.

Cannabis and cannabis-based medicines (CBM) are often used by persons with MS (PwMS).

Cannabis research to date indicates that its use worsens cognitive function in PwMS. Additionally, cognitive impairment (CI) is already a frequent consequence of MS, with a significant negative impact on quality of life (QOL).

This is pilot randomized, double blinded, double arm clinical trial of Tetrahydrocannabinol (THC) 25 mg or Cannabidiol (CBD) 50 mg orally for 15 weeks in people with MS trial.

The investigators will recruit PwMS with symptoms of neurogenic lower urinary tract dysfunction (NLUTD). These participants can either be on a treatment that has been only partially effective (as per patient report) or has never tried an intervention for their NLUTD symptoms.

The primary aim is to evaluate the differential effect of the tetrahydrocannabinol (THC) and cannabidiol (CBD) on cognitive outcomes in persons with Multiple Sclerosis (PwMS) using cannabis for NLUTD.

The results of our proposed study will better inform both healthcare practitioners and patients with respect to the potential risks of treatment with cannabis-based products and any difference with respect to THC vs. CBD-based products.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 59 years inclusive.
* Confirmed diagnosis of Multiple Sclerosis as per McDonald criteria (any type) [12]
* Symptoms of neurogenic lower urinary tract dysfunction (NLUTD) as measured by neurogenic bladder symptom score (NBSS), with a minimum score of 7.
* If already on a medication for NLUTD, must be stable on this medication for at least 4 weeks.
* Sexually active men and women of child-bearing potential must agree to use adequate contraception.
* Written informed consent.

Exclusion Criteria:

* Major psychiatric disorder such as schizophrenia or bipolar disorder
* Major neurological disorder which could affect cognition such as dementia, traumatic brain injury.
* Seizure disorder
* Use of antipsychotic medication
* Use of benzodiazepines other than exclusively at night/bedtime
* Experienced a MS relapse in the last ninety (90) days.
* Current use of cannabis or CBM greater than 3x/week.
* Currently using cannabis/CBM less than 3x/week and being unwilling to abstain for the duration of the study.
* Visual acuity (binocular) worse than 20/70 (in order to complete the cognitive outcomes)
* Significant upper extremity disability that would interfere with the cognitive tests battery.
* Indwelling catheter use/urinary diversion
* Pregnant or Breastfeeding

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Cognitive outcome: The Differential Effect, if any, of THC and CBD in MS Cognition will be measured by Symbol Digit Modality Test (SDMT). | 15 weeks
  Symbol Digit Modality Test (SDMT) is an assessment of the information processing speed. It consists of the presentation of a standard letter sized paper (8.5 × 11 in.) that contains the numbers and symbols to be processed. At the top of the page is a key where nine symbols are each paired with a single digit. The remainder of the page has a pseudorandomized sequence of these symbols. In the oral version of the SDMT, adapted for the MS population by Rao, the subject responds orally with the digit associated with each of the symbols as quickly as possible, and is scored as the total number of correct responses in 90s.Participants will be evaluated at baseline, week 10 and week 15.
NLUTD outcome: The Differential Effect, if any, of THC and CBD on Neurogenic lower urinary tract dysfunction (NLUTD) symptoms will be measured by Neurogenic Bladder Symptom Score (NBSS). | 15 weeks
  Neurogenic Bladder Symptom Score (NBSS) is a validated measure of bladder symptoms and QoL. It is scored from 0 (no symptoms) to 74 and has 3 domains: incontinence; storage, voiding, and consequences; and a single overall QOL question. Participants will be evaluated at baseline, week 10 and week 15.

SECONDARY OUTCOMES:
Blinding feasibility: The ability to blind the administration of THC vs CBD in PwMS will be evaluated based on participants and investigators report. | 15 weeks
  The investigators will ask subjects at each visit to try and identify which arm they were randomized to. If participants feel they are able to determine which group they were assigned to, they will be asked to identify how/why. This data will help investigators to develop better masking in our subsequent study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided